CLINICAL TRIAL: NCT00889122
Title: Family Exergaming: A Research Study Testing a Videogame Intervention to Increase Physical Activity for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Ann Maloney, MD, Maine Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3459
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-07

CONDITIONS: Obesity
Keywords: Obesity; Exergames; Videogames; Prevention; Family; Dance Dance Revolution; Pedometer
MeSH Terms: conditions — Obesity | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle Counseling (Experimental)
  Interventions: Behavioral: Exergame (DDR)

INTERVENTIONS:
Behavioral: Exergame (DDR) — Use of an active videogame vs. pedometers given to entire families to promote physical activity.

SUMMARY:
The purpose of this study is to determine if an interactive game (Dance Dance Revolution/DDR) can promote healthy physical activity for the health of all family members

ELIGIBILITY:
Inclusion Criteria:

* Ages 9-17
* Overweight status (BMI of 85% and above)
* Willing to come to two (2 hour) visits to MMCRI for measurements and complete surveys
* Family participation

Exclusion Criteria:

* Serious heart condition
* Photo-sensitive seizures
* Previous extensive history using DDR

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Amount of physical activity | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ann Maloney, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center Research Institute, Scarborough, Maine, United States